CLINICAL TRIAL: NCT04836533
Title: Optimizing Placebo Effects in Depressed Older Adults: Enhancing Processing Speed and Executive Functioning With Computerized Cognitive Training
Brief Title: Enhancing Processing Speed and Executive Functioning in Depressed Older Adults With Computerized Cognitive Training
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Conflicts at the study site prevented the study from being carried out
Sponsor: Queens College, The City University of New York (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); New York State Psychiatric Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: MH126187; R33MH126187 (NIH)
Record Dates: First submitted 2021-03-29; First posted 2021-04-08 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2021-03

CONDITIONS: Depression in Old Age; Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Computerized Cognitive Training (Experimental): Those assigned to the computerized cognitive training arm prior to antidepressant trial enrollment will receive computerized cognitive training that includes games that scale in difficulty.
  Interventions: Other: Experimental: Computerized Cognitive Training
- Solitaire Training (Active Comparator): Those assigned to the solitaire training arm prior to antidepressant trial enrollment will receive computerized solitaire games.
  Interventions: Other: Active Comparator: Solitaire Training
- Open-label antidepressant treatment (Experimental): Those assigned to receive open-label antidepressant treatment will begin with 10 mg of escitalopram. If the participant cannot tolerate or has an adverse reaction to escitalopram, duloxetine will be offered instead.
  Interventions: Drug: Experimental: Open-label antidepressant treatment
- Placebo-controlled antidepressant treatment (Placebo Comparator): Those assigned to the placebo-controlled group will be told that they have a 50/50 chance of receiving either escitalopram or placebo.
  Interventions: Other: Placebo Comparator: Placebo-controlled antidepressant treatment

INTERVENTIONS:
Other: Experimental: Computerized Cognitive Training — Participants will complete 4 weeks of executive functioning / processing speed training through the BrainHQ platform on their personal computers.
  Arms: Computerized Cognitive Training
Drug: Experimental: Open-label antidepressant treatment — Participants will be assigned to open-label or placebo-controlled antidepressant treatment for 8 weeks.
  Arms: Open-label antidepressant treatment
Other: Active Comparator: Solitaire Training — Participants will complete 4 weeks of Solitaire training through the BrainHQ platform on their personal computers.
  Arms: Solitaire Training
Other: Placebo Comparator: Placebo-controlled antidepressant treatment — Participants will be told they have a 50/50 chance of receiving a placebo or antidepressant.
  Arms: Placebo-controlled antidepressant treatment

SUMMARY:
The purpose of this research study is to determine how treatment response may change depending on how studies are designed, and if mobile cognitive training can be used to improve treatment response in depressed older adults.

DETAILED DESCRIPTION:
Major Depressive Disorder (MDD) is a leading cause of disability, morbidity, and mortality across the lifespan and poses a particularly severe public health problem in late life. Late-life depression (LLD) is highly recurrent, can become chronic, and is often difficult to treat. Antidepressant treatment is often ineffective in this population because of the presence of neurocognitive factors including slow processing speed (PS), executive dysfunction (ED), and cerebrovascular disease (CVD) that interfere with treatment. It is crucial, therefore, that we develop interventions that address antidepressant non-response and dramatically improve the quality of life of millions of vulnerable older adults. We recently determined that an important cause of non-response in this population is impaired expectancy effects, which in turn are compromised by slow speed of processing. We propose, therefore, that antidepressant non-response in older adults with PS deficits is caused by expectancy failure and that targeting PS deficits prior to antidepressant treatment will restore the capacity to form expectations thereby improving antidepressant treatment response. An excellent candidate for improving PS is computerized cognitive training (CCT), i.e., exercises that target, train, and strengthen specific cognitive processes with the use of structured drills and repeated practice.

To test our expectancy-processing speed model, 100 depressed adults age 60 and over with PS deficits will be recruited. Participants will be randomized to either CCT or control (Solitaire) for 4 weeks. Both conditions will train 25 minutes per day, 7 days per week. At the conclusion of this four-week period, patients will be randomly assigned to high versus low expectancy treatment conditions. Patients assigned to the low expectancy condition will be told they will receive either placebo or escitalopram when in fact they will receive escitalopram for eight weeks. Patients assigned to the high expectancy condition will be told they will receive escitalopram for eight weeks. Neuropsychological assessment will occur at baseline and weeks 4 and 12 whereas MRI scans will be conducted at baseline and week 4.

Clinical assessments will be conducted biweekly throughout the study. The goals of this study are to 1) To determine whether PS mediates the relationship between CCT and expectancy, and 2) To compare endpoint depression scores as a function of CCT and expectancy conditions.

At the screening evaluation, informed consent for the screening evaluation is obtained. Participants subsequently undergo a psychiatric clinical interview using the Structured Clinical Interview Diagnostic for DSM-V (SCID-V), 24- item Hamilton Rating Scale for Depression (HRSD), Clinical Global Impressions Scale - Severity (CGI-Severity), Cumulative Illness Rating Scale for Geriatrics (CIRS-G) and Antidepressant Treatment History Form (ATHF) to document depression diagnosis, severity, and medical comorbidity. WAIS-IV Digit Symbol Coding will be completed to determine whether the patient meets inclusion criteria for PS (>1 SD on age adjusted norms). If the patient is eligible for study entry, participation in the research protocol will be discussed and informed consent will be obtained. After consent is obtained, patients will receive a comprehensive baseline neuropsychological assessment and MRI (structural, resting state, and DTI). Neuropsychological assessments include MMSE, WAIS-IV Coding, NIH Toolbox Cognition Battery, NIH Supplement Auditory Verbal Learning Test (Rey), Trail Making Test (Part A and B), Stroop Color-Word Test, and The Letter and Animal Naming Test. These measures will capture global cognitive functioning, processing speed, attention, and response inhibition, and verbal fluency. After testing, patients will be randomized to either CCT or active control for 4 weeks (25'/day, 7 days/week). Patients randomized to CCT will complete seven 25-minute sessions per week for 4 weeks using BrainHQ's Double Decision in the experimental condition (a processing speed exercise) and BrainHQ solitaire in the control condition. At the conclusion of this four-week period, patients will complete a second neuropsychological assessment and a second fMRI (to determine change in resting-state BOLD signal in the CCN). Patients will then be randomly assigned to high versus low expectancy treatment conditions. Patients assigned to the low expectancy condition will be told they will receive either placebo escitalopram when in fact they will receive escitalopram for eight weeks. Patient assigned to the high expectancy condition will be told and they will receive escitalopram for eight weeks. Expectancy is measured at baseline and after informing patients of their randomization status. The difference between their pre and post randomization expectancy regarding treatment improvement is the expectancy effect. At the conclusion of the eight-week clinical trial, the difference in antidepressant response observed between the open and placebo-controlled medication treatments is a measure of the expectancy contribution to outcome. Neuropsychological assessment will occur again at the conclusion of the escitalopram trial (week 12). Clinical assessments will be conducted biweekly throughout the study.

The novel experimental therapeutics approach taken in this proposal cuts across several research themes (prevention and translation) and addresses many of the challenges (digital technology and neural circuits) elaborated in NIMH's Strategic Plan for mental health research in the 21st century. Consistent with NIMH goals, it also develops strategies for tailoring existing interventions to optimize outcomes and elucidates the mechanism by which antidepressant treatment in LLD can be restored.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than or equal to 60 years
2. DSM5 Diagnosis of Major Depressive Disorder (MDD), Persistent Depressive Disorder, or Depression Not Otherwise Specified (NOS)
3. Hamilton Rating Scale for Depression (HRSD) score ≥ 20
4. Decreased processing speed (1 SD below age-adjusted norms on the WAIS-IV Digit Symbol Coding Test)
5. Access to a computer with daily internet access
6. Willing to and capable of providing informed consent and complying with all study procedures. At the end of the CCT phase (week 4), depression severity will be reassessed. To be eligible for Phase 2 (SSRI trial), participants will be required to have an HRSD score ≥ 14.

Exclusion Criteria:

1. Diagnosis of substance abuse or dependence (excluding Tobacco Use Disorder) within the past 12 months
2. History of psychosis, psychotic disorder, mania, or bipolar disorder
3. Primary neurological disorder, including dementia, stroke, Parkinson's disease, epilepsy, etc.
4. Mini Mental Status Examination (MMSE) score less than 24
5. HRSD suicide item greater than 2 or Clinical Global Impressions (CGI)-Severity score of 7 at baseline
6. History of allergic or adverse reaction to escitalopram, or non-response to adequate trial of escitalopram (at least 4 weeks at dose of 20 mg) during the current episode
7. Current or recent (within the past 2 weeks) treatment with psychotherapy, antidepressants, antipsychotics, mood stabilizers
8. Contraindication to MRI scanning (such as metal in body) or inability to tolerate the scanning procedures
9. History of significant radioactivity exposure (nuclear medicine studies or occupational exposure).

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01-31 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Hamilton Rating Scale for Depression (HRSD) Change | Screen, Weeks 0, 1, 2, 3, 4, 6, 8, 10, 12
  Clinician-rated measure of depressive severity composed of 24 questions used to measure changes in depressive symptoms and monitor safety during the study.
Treatment Credibility Expectancy Scale (CES) - item 4 Change | Baseline, Week 0
  Self-report scale in which subjects rate their impression of the credibility of the treatment and how they estimate their expectation of improvement. Item 4 measures how much improvement in depression symptoms is expected.
Processing Speed Change - WAIS-IV Coding | Baseline, Weeks 4, 12
  Processing speed will be assessed using Coding from the Wechsler Adult Intelligence Scale-IV (WAIS-IV), the NIH Toolbox Pattern Comparison Processing Speed Test, and Trail Making Test A. From these 3 tests, a composite score (primary outcome) is derived by extracting a latent factor and factor loadings, creating a purer measure of processing speed than raw scores from an individual test or a sum total score.
Processing Speed Change - NIHH Toolbox Pattern Comparison Processing Speed Test | Baseline, Weeks 4, 12
  Processing speed will be assessed using Coding from the Wechsler Adult Intelligence Scale-IV (WAIS-IV), the NIH Toolbox Pattern Comparison Processing Speed Test, and Trail Making Test A. From these 3 tests, a composite score (primary outcome) is derived by extracting a latent factor and factor loadings, creating a purer measure of processing speed than raw scores from an individual test or a sum total score.
Processing Speed Change - Trail Making Test A | Baseline, Weeks 4, 12
  Processing speed will be assessed using Coding from the Wechsler Adult Intelligence Scale-IV (WAIS-IV), the NIH Toolbox Pattern Comparison Processing Speed Test, and Trail Making Test A. From these 3 tests, a composite score (primary outcome) is derived by extracting a latent factor and factor loadings, creating a purer measure of processing speed than raw scores from an individual test or a sum total score.
Resting State Functional Connectivity Index Change | Baseline, Week 4
  Measure of resting state fMRI.

SECONDARY OUTCOMES:
Secondary Clinical Global Impressions (CGI) Severity and Improvement | Screen, Weeks 0, 1, 2, 3, 4, 6, 8, 10, 12
  Scales measuring the clinician's view of subjects' global functioning that will provide a clinical assessment of subjects at each visit and help maintain safety by identifying clinical worsening.
Inventory for Depressive Symptomatology Self-Report (IDS-SR) | Weeks 0, 1, 2, 3, 4, 6, 8, 10, 12
  The IDS-SR is a standard self-report measure of depression severity that will be used to measure changes in depressive symptoms and monitor safety during the study.
Cumulative Illness Rating Scale for Geriatrics (CIRS-G) | Screen
  Provides quantitative ratings of chronic illness burden. Presence of illness is rated from 0 to 4 in 14 different medical domains. Scores range from 0-56.
NIH Toolbox Auditory Verbal Learning Test - Rey (RAVLT) | Baseline, Weeks 4, 12
  Measures immediate recall. Unrelated words presented via audio recording and participant recalls as many as possible
Stroop Color-Word Test (Stroop) | Measure of response inhibition sensitive to frontal lobe dysfunction. This test is divided into three conditions: color naming, word reading, and colorword inhibition.
  Baseline, Weeks 4, 12
Letter and Animal Naming Test | Baseline, Weeks 4, 12
  Test measuring the verbal fluency component of executive functioning. Requires subjects to generate words that begin with a particular letter or belong to a particular semantic category as quickly as possible
World Health Organization Disability Assessment Schedule 2.0 (WHODAS2.0) | Screen, Weeks 4, 6, 8, 10, 12
  This 36-item self-report provides a global measure of disability and 7 domain-specific scores based on the conceptual framework of the International Classification of Functioning, Disability, and Health (ICF).
Trail Making Test A and B | Baseline, Weeks 4, 12
  Paper and pencil test that assesses (A) speeded attention and (B) the switching component of executive function. This test has two conditions: (A) number sequencing and (B) number-letter sequencing.
NIH Toolbox Flanker Inhibitory Control and Attention Test | Baseline, Weeks 4, 12
  Measures attention and executive functioning. The allocation of one's limited capacities to deal with an abundance of environmental stimulation
NIH Toolbox Picture Sequence Memory Test | Baseline, Weeks 4, 12
  Measures episodic memory. Cognitive processes involved in the acquisition, storage, and retrieval of new information.
NIH Toolbox List Sorting Working Memory Test | Baseline, Weeks 4, 12
  Measures working memory. The ability to store information until the amount of information to be stored exceeds one's capacity to hold that information.
NIH Toolbox Picture Vocabulary Test | Baseline, Weeks 4, 12
  Measures receptive vocabulary administered in a computer-adaptive test (CAT) format. Respondents select the picture that most closely matches the meaning of the word.
NIH Toolbox Oral Reading Recognition Test | Baseline, Weeks 4, 12
  Measures reading and decoding skill and crystallized abilities. Participant is asked to read and pronounce letters and words as accurately as possible.
NIH Toolbox Dimensional Card Change Sort Test | Baseline, Weeks 4, 12
  Measures executive function. The capacity to plan, organize and monitor the executive of behaviors that are strategically directed in a goal-oriented manner.
NIH Toolbox Pattern Comparison Processing Speed Test | Baseline, Weeks 4, 12
  Assesses the amount of information that can be processed within a certain unit of time. Items are simple so as to purely measure processing speed.
Diffusion Tensor Imaging (fractional anisotropy and mean diffusivity) | Baseline, Week 4
  Measures of brain white matter integrity.

OTHER OUTCOMES:
Structured Clinical Interview Diagnostic for DSM-V (SCIDV) | Screen
  Structured clinical interview to assess current and past psychiatric diagnoses.
Mini-Mental Status Exam (MMSE) | Screen
  A brief, structured 30-item mental status examination that measures concentration or working memory, language and praxis, orientation, memory, and attention span
Wechsler Adult Intelligence Scale-IV (WAIS-IV) Digit Symbol Coding | Screen, Weeks 4, 12
  Participants are required to copy symbols paired with numbers in a 120 second time limit. The score is the number correct in the allotted time.

CONTACTS AND LOCATIONS:
Overall Officials: Joel R Sneed, PhD, Principal Investigator — Queens College and NYSPI
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No